CLINICAL TRIAL: NCT00483197
Title: Evaluation of the VentrAssistTM Left Ventricular Assist Device as a Bridge to Cardiac Transplantation - Pivotal Trial
Brief Title: VentrAssistTM LVAD as a Bridge to Cardiac Transplantation - Pivotal Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ventracor (Industry)
Collaborators: International Center for Health Outcomes and Innovation Research (Other)
Responsible Party: Nader Moazami, MD Sugical PI, Washington Hospital/Barnes Jewish Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP 06005
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: End-stage Heart Failure; Cardiomyopathies
Keywords: VentrAssistTM; LVAD; End-stage heart failure; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: VentrAssistTM Left Ventricular Assist Device

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of VentrAssistTM LVAD in individuals who are awaiting heart transplants.

DETAILED DESCRIPTION:
LVADs are efficacious in improving survival and functional status when used as a bridge to transplantation. The purpose of this study is to evaluate the safety and effectiveness of the VentrAssist LVAD in providing circulatory support in individuals who are awaiting heart transplants.

The VentrAssist LVAD is a centrifugal flow pump. Its small size and mechanical simplicity offers benefits not available with currently approved LVADs, including facilitating a more limited implantation procedure, which could reduce surgical morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:(The following are general criteria; more specific criteria are included in the study protocol):

* Approved and listed for cardiac transplantation.
* Patient for whom LVAD implantation is planned as a clinically indicated bridge to cardiac transplantation.

Exclusion Criteria:(The following are general criteria; more specific criteria are included in the study protocol):

* Presence of heart conditions that would contraindicate LVAD implantation by adversely affecting patient survival or LVAD function.
* Primary coagulopathy or platelet disorder; contraindication to anticoagulant or anti-platelet agents.
* Presence of any mechanical circulatory support other than intra-aortic balloon pump.
* Therapy with an investigational intervention at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-06; Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Survival to cardiac transplantation or to 180 days post implantation and listed for cardiac transplantation in categories UNOS 1A or 1B.

SECONDARY OUTCOMES:
Quality of life
Functional status
Neurocognitive function

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - University of Florida, Gainesville, Florida
  - Jackson Memorial, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St. Vincent's, Indianapolis, Indiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Columbia University, New York, New York
  - Rochester Medical Center University, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Fairfax (Inova) Hospital, Falls Church, Virginia
  - University of Washington, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin Hospital, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin